CLINICAL TRIAL: NCT04194047
Title: Effects of Red Blood Cells Transfusion on Renal Resistivity Index and Renal Venous Stasis Index
Brief Title: Effects of Red Blood Cells Transfusion on Renal Blood Flow
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Fogagnolo, Principal Investigator, Università degli Studi di Ferrara
Other Study IDs: RRIRBC
Record Dates: First submitted 2019-12-08; First posted 2019-12-11 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Acute Kidney Injury; Transfusion-Associated Circulatory Overload; Anemia; Fluid Overload
MeSH Terms: conditions — Acute Kidney Injury; Transfusion Reaction; Anemia; Edema | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RBC group: Patients who received RBC transfusion
  Interventions: Other: Transfusion
- crystalloids group: Patients who received fluid resuscitation with crystalloids
  Interventions: Other: Crystalloids infusion
- control group: Patients not receiving RBC nor crystalloids

INTERVENTIONS:
Other: Transfusion — RBC transfusion (1 unit)
  Groups: RBC group
Other: Crystalloids infusion — Infusion of 500 ml of balanced crystalloids
  Groups: crystalloids group

SUMMARY:
The renal Doppler resistive index (RRI) is a noninvasive tool that has been used to assess renal perfusion in the intensive care unit (ICU) setting. It is associated with the occurrence of acute kidney injury (AKI). Many parameters have been described as influential on the values of renal RI. Red blood cell (RBC) transfusion were shown to be able to increase renal oxygenation in animal model, whereas crystalloid resuscitation did not. We sought to describe the different effect of crystalloids infusion and RBC transfusion on renal blood flow, as evaluated with doppler ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 90
* Hemoglobin ≥7 and ≤ 10 g/dl

Exclusion Criteria:

* Ultrasound RRI evaluation non available
* Patients with arrhythmia
* Pregnancy
* Refusal to give consent
* History of renal transplantation
* Central venous access in superior vena cava not available Critical active bleeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of critically ill patients
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in renal resistivity index (RRI) after intervention | after 60 minute from intervention
  To compare change in RRI after intervention between groups. Values over>0.70 are considered pathological. Higher values means worse outcome.
Change Renal Venous Stasis Index (RSVI) after intervention | after 60 minute from intervention
  To compare change in RSVI after intervention between groups. Under physiological conditions, the index is zero. Higher values means worse outcome.

SECONDARY OUTCOMES:
Occurence of AKI | Once a day for 7 days
  Occurence of AKI as defined by Kidney Disease: Improving Global Outcomes (KDIGO)
Variation in renal resistivity index (RRI) | after 24 hours from intervention
  To compare change in RRI after intervention between groupsValues over>0.70 are considered pathological. Higher values means worse outcome.
Variation in Renal Venous Stasis Index (RSVI) | after 24 hours from intervention
  To compare change in RSVI after intervention between groups. Under physiological conditions, the index is zero. Higher values means worse outcome.

OTHER OUTCOMES:
correlation between arterial-venous oxygen differences and changes in renal resistivity index (RRI) after intervention | after 24 hours from intervention
  RRI values over>0.70 are considered pathological. Higher values means worse outcome.
correlation between arterial-venous oxygen differences and changes in Renal Venous Stasis Index (RSVI) | after 24 hours from intervention
  Under physiological conditions, the index is zero. Higher values means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zafrani L, Ergin B, Kapucu A, Ince C. Blood transfusion improves renal oxygenation and renal function in sepsis-induced acute kidney injury in rats. Crit Care. 2016 Dec 20;20(1):406. doi: 10.1186/s13054-016-1581-1. PMID 27993148
- [Background] Husain-Syed F, Birk HW, Ronco C, Schormann T, Tello K, Richter MJ, Wilhelm J, Sommer N, Steyerberg E, Bauer P, Walmrath HD, Seeger W, McCullough PA, Gall H, Ghofrani HA. Doppler-Derived Renal Venous Stasis Index in the Prognosis of Right Heart Failure. J Am Heart Assoc. 2019 Nov 5;8(21):e013584. doi: 10.1161/JAHA.119.013584. Epub 2019 Oct 19. PMID 31630601